CLINICAL TRIAL: NCT06959160
Title: Comparison of the Immediate Effects of Manual Therapy Techniques on Joint Range of Motion, Grip Strength, Pressure Pain Threshold, and Functionality in Non-Specific Neck Pain
Brief Title: Comparison of the Immediate Effects of Manual Therapy Techniques in Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acetinkaya006
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Manual Therapies; Neck Pain
Keywords: Manual Therapy Techniques; Non-Specific Neck Pain; Immediate Effects
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atlanto-occipital Manipulation Group (Experimental): Participants in the first group received atlanto-occipital manipulation.
  Interventions: Other: Atlanto-occipital manipulation
- Cervical Mobilization Group (Experimental): Participants in the second group underwent Grade II-III cervical mobilization techniques.
  Interventions: Other: Cervical mobilization
- Trigger Point Therapy Group (Experimental): Participants in the third group received trigger point therapy, which included ischemic compression followed by myofascial stretching on the upper trapezius muscle.
  Interventions: Other: Trigger point therapy

INTERVENTIONS:
Other: Atlanto-occipital manipulation — Participants in the first group received atlanto-occipital manipulation. The patient was positioned in a supine position, with the head rotated to one side. The therapist placed the middle and ring fingers of one hand on the patient's mastoid process, while the palm of the other hand made contact with the patient's jawline and cheek. A gentle traction force was applied to the cranial region using both hands. When the therapist sensed joint tension, a high-velocity, low-amplitude thrust was delivered in the direction of the traction with a slight rotational force. The procedure was performed bilaterally and lasted approximately 5 minutes.
  Arms: Atlanto-occipital Manipulation Group
Other: Cervical mobilization — Participants in the second group underwent Grade II-III cervical mobilization techniques, administered over a period of 10 minutes. The patient was positioned in a supine position, and the physiotherapist performed 10 minutes of Grade II-III mobilizations with an upward and downward incline (postero-anterior and antero-posterior mobilizations following the movement plane of the cervical zygapophyseal joints).
  Arms: Cervical Mobilization Group
Other: Trigger point therapy — Participants in the third group received trigger point therapy, which included ischemic compression followed by myofascial stretching on the upper trapezius muscle. The patient was positioned in a supine position, and the physiotherapist performed 10 minutes of Grade II-III mobilizations with an upward and downward incline (postero-anterior and antero-posterior mobilizations following the movement plane of the cervical zygapophyseal joints).
  Arms: Trigger Point Therapy Group

SUMMARY:
The aim of this study is to investigate the effects of manual therapy techniques on joint range of motion, pain tolerance, grip strength, and functionality in individuals with non-specific neck pain. The study is experimental in design. Individuals aged between 18 and 55 who were diagnosed with non-specific neck pain and met the inclusion criteria participated in the study.

DETAILED DESCRIPTION:
Participants who agreed to take part and signed the informed consent form were asked to complete the "Patient Assessment Form" during the initial interview.

In addition, the following assessment tools were used: the Cervical Range of Motion (CROM) device to evaluate joint range of motion, a hand dynamometer to assess grip strength, an algometer to measure pain tolerance, and the "Neck Disability Index" to evaluate functionality.

Participants were then randomly assigned to one of three groups:

Group 1: Atlanto-occipital manipulation

Group 2: Cervical mobilization

Group 3: Trigger point therapy

Participants in the first group received atlanto-occipital manipulation, those in the second group underwent Grade II-III mobilization techniques, and those in the third group received trigger point therapy, which consisted of ischemic compression followed by myofascial stretching on the upper trapezius muscle.

Immediately after the treatments, joint range of motion, pain tolerance, and functionality were reassessed. The manual therapy interventions for all three groups were performed by different specialized physiotherapists trained in these techniques. The evaluations, however, were conducted by another physiotherapist who was blinded to the treatments (double-blind study).

The data were statistically analyzed using the Statistical Package for the Social Sciences program, and a p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 55
* Have been diagnosed with non-specific neck pain by a specialized physician
* Have been experiencing neck pain for less than 3 months
* Have a neck pain level of at least 3 on the Visual Analog Scale
* Have bilateral active trigger points in the upper trapezius muscle
* Have restricted active cervical range of motion

Exclusion Criteria:

* Presence of neurological deficit or radicular pain
* History of pathology or surgery in the cranio-cervical region
* Positive response in the extension-rotation test
* Use of anticoagulants or corticosteroids
* Presence of one or more red flags defined for non-specific neck pain

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Cervical Joint Range of Motion | Immediately before and after interventions, assessed within a single session
  The evaluation of cervical flexion, extension, right-left lateral flexion, and right-left rotation range of motion conducted using the CROM device. The CROM device is an inclinometer system affected by magnetic forces and gravity. Validity and reliability studies have been carried out to assess the movements of the cervical region using this device. There are no risks or side effects associated with this assessment method.
Assessment of Grip Strength | Immediately before and after interventions, assessed within a single session
  Grip strength of the individuals was measured using the "Jamar Hand Dynamometer" (Takei Scientific Instruments Co., Ltd. - Japan). Measurements were conducted as recommended in the literature, with the patient comfortably seated, shoulder abducted, elbow in 90 degrees of flexion, forearm in a neutral position, and wrist in 0-30 degrees of extension. Measurements were repeated three times with five-second intervals between each trial for both the dominant and non-dominant hands, and the average value was recorded as the result. There are no risks or side effects associated with this assessment method.
Measurement of Pain Tolerance Threshold | Immediately before and after interventions, assessed within a single session
  Pain tolerance was measured using the J-tech algometer device. Measurements were taken bilaterally, both on the right and left sides, at the C5 level and at the midpoint of the upper trapezius muscle. The measurements were repeated three times, and the average value was recorded as the result. There are no risks or side effects associated with this assessment method.
Neck Disability Index | Immediately before and after interventions, assessed within a single session
  This questionnaire is used for the evaluation of cervical function and has undergone validity and reliability studies. The questionnaire consists of 10 sections, with 6 multiple-choice options for each section. Scoring ranges from 0 to 5 for each section based on the selected response. The total score determines the overall result of the test. There are no risks or side effects associated with this assessment method.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, assoc. prof., Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No